CLINICAL TRIAL: NCT05186896
Title: NETTUNIT - Italy-Tunisia Cross-border Environmental network_2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Responsible Party: Principal Investigator, Stefania La Grutta, MD, Research Director, Istituto per la Ricerca e l'Innovazione Biomedica
Other Study IDs: 03/2021_2
Record Dates: First submitted 2021-11-16; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Risk Perception

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Residents of areas at high risk of environmental crisis: 1000 adult males and females living in areas declared at high risk of environmental crisis in the areas of Caltanissetta (Italy) and Tunis (Tunisia).
  Interventions: Other: Risk perception questionnaire

INTERVENTIONS:
Other: Risk perception questionnaire — A questionnaire for risk perception will be developed and administered

SUMMARY:
The study involves the development and validation of a questionnaire for risk perception to be administered to residents of areas declared to be at high risk of environmental crisis in the areas of Caltanissetta (Italy) and Tunis (Tunisia). The questionnaire will be administered twice, at baseline and after 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 20-90 years of both sex, living in the areas of Caltanissetta (Italy) and Tunis (Tunisia).

Exclusion Criteria:

* Individuals with learning difficulties.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals aged 20-90 years of both sex, living in the areas of Caltanissetta (Italy) and Tunis (Tunisia).
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-03-03 (Estimated); Study Completion 2023-03-03 (Estimated)

PRIMARY OUTCOMES:
Construct validity of the questionnaire score at baseline administration | Baseline administration
  The ability of the questionnaire score at baseline to differentiate between sub-samples that are known or expected to differ
Construct validity of the questionnaire score 1 month after the baseline administration | 1 month after the baseline administration
  The ability of the questionnaire score 1 month after the baseline administration to differentiate between sub-samples that are known or expected to differ
Repeatability of the questionnaire score between the first (baseline) and second (1 month) administration | Baseline administration and 1 month after the baseline administration
  The extent to which the answer distribution will be similar between the two administrations

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR), Palermo, Italy